CLINICAL TRIAL: NCT01704820
Title: RIGHT SIDED COLON POLYP MISS RATE: IMPACT OF RETROFLEXION IN THE RIGHT COLON
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Washington University School of Medicine (Other)
Collaborators: Medical College of Wisconsin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: Retro-View
Record Dates: First submitted 2012-10-08; First posted 2012-10-11 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: Colon Polyps; Colon Cancer Screening
Keywords: Colon Polyps; Colon Cancer screening; Colonoscopy
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Retroflexion arm (Experimental): Retroflexion arm: retroflexion in the cecum or proximal ascending colon and slow withdrawal to the hepatic flexure with removal of all visible colon polyps
  Interventions: Procedure: Retroflexion in the right colon
- Forward view arm (Placebo Comparator): Colonoscope is slowly withdrawn from the proximal colon to the hepatic flexure and all visible colon polyps are removed.

INTERVENTIONS:
Procedure: Retroflexion in the right colon
  Arms: Retroflexion arm

SUMMARY:
Colonoscopy is the gold standard screening test for colorectal cancer. Removal of pre-malignant colon polyps during colonoscopy reduces colorectal cancer mortality by over 50%. However, while colonoscopy is highly effective at preventing distal (left sided) colon cancers, it provides only limited protection from cancer in the proximal (right side) colon. Our goal is to determine if additional pre-cancerous colon polyps can be identified by looking at the right side of the colon in retroflexion. During retroflexion the tip of the colonoscope is turned 180 degrees; allowing the doctor to view the backs of colonic folds. If additional polyps can be identified in this manner colonoscopy will become a more efficient method of screening for colon cancer.

In order to evaluate how effective right colon retroflexion is at detecting polyps in the proximal colon we plan on performing a randomized, controlled trial. Patients undergoing screening or follow up colonoscopy will be invited to participate in the study. Those patients who agree to participate will be randomized into one of two groups once the colonoscope is fully inserted. Group one will have the right side of their colon examined for polyps with the endoscope looking forward (traditional form of examination) followed by repeat examination of the right side of the colon with the colonosocpe in retroflexion (looking backwards). Polyps seen during each section of the exam will be removed and manner in which the polyps were found/ removed will be recorded. Following the two exams of the right side of the colon the colonoscopy will be completed in the usual manner. The duration of each portion of colonoscopy will be recorded. After the procedure is completed the physician performing the colonoscopy will rate difficulty of the procedure and confidence with quality of the examination. Pathology results for each polyp will be recorded once available. There will be no study related follow up after the pathology results are recorded.

ELIGIBILITY:
Inclusion Criteria:

* • Patients >18 years of age undergoing colonoscopy for colorectal cancer screening or routine polyp surveillance

Exclusion Criteria:

* • Failure to intubate the cecum during colonoscope insertion

  * Prior right colon resection
  * Known polyposis syndrome or polyposis identified at colonoscopy
  * Inflammatory bowel disease
  * Preparation of the colon is judged fair or poor using Boston Bowel Preparation Scale.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1020 (Estimated)
Dates: Start 2012-09; Primary Completion 2014-09 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Per patient adenoma detection rate (average # adenomas detected/ patient in each arm of the study). | 2 weeks
  The primary objective of our study is to determine whether the diagnostic yield for pre-malignant polyps is increased by retroflexion of the colonoscope during withdrawal from the proximal colon when compared to the diagnostic yield of a second examination of the proximal colon with the colonoscope in forward view.

SECONDARY OUTCOMES:
Evaluate the success rate of retroflexion in the proximal colon. | 1 day
  Evaluate the percent of patients in whom retroflexion can be performed.
Identify risk factors for missing polyps on first examination of right colon | 1 day
  We will perform a multivariable analysis in order to identify patient and procedure related factors which are associated with missed polyps.
Access whether duration of exam is different in the retroflexion vs. forward view arms of the study. | 1 day
  Access whether duration of exam is different in the retroflexion vs. forward view arms of the study. By timing all portions of the exam.
Evaluate endoscopist comfort with performing retroflexion in the proximal colon. | 1 day
  Evaluate endoscopist comfort with performing retroflexion in the proximal colon using a 5 point Likert scale

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Washington University in St Louis, St Louis, Missouri
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Background] Hewett DG, Rex DK. Miss rate of right-sided colon examination during colonoscopy defined by retroflexion: an observational study. Gastrointest Endosc. 2011 Aug;74(2):246-52. doi: 10.1016/j.gie.2011.04.005. Epub 2011 Jun 15. PMID 21679946